CLINICAL TRIAL: NCT02526420
Title: An Open-Label, Dose Finding, International Phase 2 Study With Once Monthly Subcutaneous VRS-317 in Adult Growth Hormone Deficiency (GHD)
Brief Title: Versartis International Trial in Adults With Long-Acting Growth Hormone
Acronym: VITAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Versartis Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Organization: Aravive, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15VR7
Record Dates: First submitted 2015-08-13; First posted 2015-08-18 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Adult Growth Hormone Deficiency
Keywords: VRS-317; Long Acting Growth Hormone; Versartis; somavaratan; Growth Hormone Deficiency; Adult Growth Hormone Deficiency; AGHD; Growth Hormone Replacement; Growth Hormone Replacement Therapy; XTEN
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort A: Somavaratan in Older Adults (Experimental): Long-acting recombinant human growth hormone therapy administered subcutaneously once monthly in subjects >= 35 years of age
  Interventions: Drug: somavaratan
- Cohort B: Somavaratan in Younger Adults (Experimental): Long-acting recombinant human growth hormone therapy administered subcutaneously once monthly in subjects < 35 years of age
  Interventions: Drug: somavaratan
- Cohort C: Somavaratan in Women on Estrogen (Experimental): Long-acting recombinant human growth hormone therapy administered subcutaneously once monthly in female subjects on oral estrogen (regardless of age)
  Interventions: Drug: somavaratan

INTERVENTIONS:
Drug: somavaratan — Long-acting recombinant human growth hormone therapy administered subcutaneously once monthly
  Other Names: VRS-317

SUMMARY:
A Phase 2, open-label dose-finding safety study of individualized monthly VRS-317 dosing for five months in adults with GHD.

DETAILED DESCRIPTION:
A Phase 2, dose finding safety study to evaluate an individualized monthly VRS-317 dosing regimen in adults with GHD. This is an open-label, international, multicenter study with VRS-317 treatment for five months. This treatment period will include monthly dose titrations until a subject's mean IGF-I SDS value is within a target range for two consecutive months. Subjects will be stratified into three cohorts based on sensitivity to rhGH.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of childbearing potential must have negative pregnancy test and use appropriate contraceptive methods
* Subjects must have documented GHD during adulthood.
* Subjects taking other hormone replacement therapy must have been on a stable course of treatment for at least 3 months.
* Subjects with underlying disorders responsible for the subject's GHD must have been clinically stable for at least 6 months.
* Subjects receiving daily rhGH injections must washout for 14 days.
* Subjects must provide signed informed consent.
* Subjects must have a BMI (kg/m2) between 19.0 and 35.0.

Exclusion Criteria:

* Subjects with diabetes mellitus or inadequate glucose control
* Subjects with untreated adrenal insufficiency.
* Subjects with free thyroxine outside the normal reference range.
* Subjects currently taking oral glucocorticoids, except for physiological maintenance doses of oral glucocorticoids in subjects with multiple pituitary hormone deficiencies.
* Subjects with current significant cardiovascular disease, heart insufficiency of NYHA class > 2.
* Subjects with current significant cerebrovascular, pulmonary, neurological, renal, inflammatory, or hepatobiliary disease.
* Subjects with current papilledema.
* Subjects with a history of persistent or recurring migraines.
* Subjects with current edema (≥ CTCAE Grade 2).
* Subjects with current drug or alcohol abuse.
* Subjects with a documented history of HIV, current HBV or HCV infection
* Subjects with a prior history of malignancy excluding adequately treated non-melanoma skin cancers or in situ carcinoma of the cervix.
* Women who are pregnant or breastfeeding.
* Subjects with a significant abnormality in Screening laboratory results

Ages: 23 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Safety as measured by the number of subjects with adverse events, concomitant medications, safety labs, vital signs and physical exams | 5 months
  Safety observations include adverse events, concomitant medications, safety labs, vital signs and physical exams.
Starting doses (proportion of subjects who achieve normalization of IGF-I SDS response during the first dosing interval ) | 5 months
  To evaluate the starting doses of VRS-317 for each cohort as measured by the proportion of subjects who achieve normalization of IGF-I SDS response during the first dosing interval (one month after the first dose)
Dose titration plan (proportion of subjects who achieve a mean IGF-I SDS within the defined target range after each dose titration) | 5 months
  To evaluate the dose titration plan of VRS-317 for each cohort as measured by the proportion of subjects who achieve a mean IGF-I SDS within the defined target range after each dose titration

SECONDARY OUTCOMES:
Immunogenicity of VRS-317 by measurement of serum anti-drug antibody (ADA) titers | 5 months
  To evaluate the immunogenicity of VRS-317 by measurement of serum anti-drug antibody (ADA) titers
Immunogenicity of VRS-317 by detection of neutralizing antibodies (NAbs) | 5 months
  To evaluate the immunogenicity of VRS-317 by detection of neutralizing antibodies (NAb)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Rogoff, MD, PhD, Study Director — Versartis Inc.
Locations (18):
- United States (9):
  - AMCR Institute Inc., Escondido, California
  - Therapeutic Research Institute of Orange County, Laguna Hills, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Palm Research Center, Las Vegas, Nevada
  - Endocrine Associates of Dallas, Plano, Texas
  - Swedish Medical Center, Seattle, Washington
- Australia (3):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - St Vincent's Hospital, Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Germany (2):
  - Charite-Universitätsmedizin, Berlin
  - Universitätsklinikum Essen, Essen
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham, B152gw
  - William Harvey Research Institute, London, EC1M 6BQ
  - Hull Royal Infirmary, Hull, East Yorkshire, HU3 2RW
  - The Christie NHS Foundation Trust, Manchester, M20 4BX

REFERENCES:
- See also: Company Website — http://www.versartis.com